CLINICAL TRIAL: NCT05029765
Title: A 24 Weeks Double-blind Latin-square Trial of Effect of Mediterranean Diet and Probiotics in Adults With Mild Cognitive Impairment
Brief Title: Effect of Mediterranean Diet and Probiotics in Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pablo Pérez Martínez (Other)
Responsible Party: Sponsor-Investigator, Pablo Pérez Martínez, Investigator-in-charge at Nutrigenomics Metabolic Syndrome group, Maimónides Biomedical Research Institute of Córdoba
Organization: Maimónides Biomedical Research Institute of Córdoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PI16/01777
Record Dates: First submitted 2018-06-14; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Probiotics; Microbiota; Mediterranean diet
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Diet, Mediterranean; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: 50 men and women with mild cognitive impairment and more than 60 years will follow three dietary intervention periods of 24 weeks each, with a randomized crossover design. Dietary periods will be: 1.- Healthy diet (WHO recommendations) + placebo; 2.- Mediterranean diet + placebo and ; 3.- Mediterranean diet "plus" (Mediterranean diet + Biopolis-MIX42 (a capsule containing 10^9 colony forming units of Lactobacillus rhamnosus and Bifidobacterium longum)).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy diet Arm (Placebo Comparator): Healthy diet (WHO recommendations) + placebo
  Interventions: Dietary Supplement: Healthy diet (WHO recommendations); Dietary Supplement: Placebo
- Mediterranean diet Arm (Placebo Comparator): Mediterranean diet + placebo
  Interventions: Dietary Supplement: Mediterranean diet; Dietary Supplement: Placebo
- Mediterranean diet "plus" Arm (Active Comparator): Mediterranean diet + Biopolis-MIX42 (1 capsule per day containing 10^9 colony forming units of Lactobacillus rhamnosus and Bifidobacterium long).
  Interventions: Dietary Supplement: Mediterranean diet; Dietary Supplement: Biopolis-MIX42

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — Mediterranean diet:
  22% Monounsaturated fat, 6% Polyunsaturated fat, 7% Saturated fat, 15% Protein, 50% Carbohydrates
  Arms: Mediterranean diet "plus" Arm; Mediterranean diet Arm
Dietary Supplement: Healthy diet (WHO recommendations) — Recommendations according to WHO
  Arms: Healthy diet Arm
Dietary Supplement: Placebo — Placebo
  Arms: Healthy diet Arm; Mediterranean diet Arm
Dietary Supplement: Biopolis-MIX42 — Biopolis-MIX42: a capsule containing 10^9 colony forming units of Lactobacillus rhamnosus and Bifidobacterium longum.
  Arms: Mediterranean diet "plus" Arm

SUMMARY:
Manipulation of the gut microbiota through dietary modification affects brain function, with improvement in patients with cognitive disorders. Combined effect of nutritional intervention with Mediterranean diet and probiotics with potentially healthy growth of germ, affect the evolution of mild cognitive impairment, by the modulation of components related with the axis microbiota-gut-brain: neuropeptides, short-chain fatty acids, markers for oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 60 years with mild cognitive impairment (Clinical Dementia Rating (CRD) 0.5; Mini Mental Examiantion de Folstein (MMSE)> 23; Repeatable Battery for the Asessment of Neuropsychological Status (RBANS) <= 85)
* Drugs with a stable dose from a minimum of 4 weeks prior to screening (excluding psychopharmaceuticals and any other that could affect alertness and cognitive ability)
* Geriatric depression scale score <6
* Sufficient visual and auditory abilities to carry out the neuropsychological tests. Good health without diseases that prevent the completion of the study.
* A minimum educational training established for 6 years or similar work history.
* A familiar informant or close caregiver with a minimum contact with the patient established in 10 hours per week that can accompany the participant to the clinical visits

Exclusion Criteria:

* Any uncontrolled medical or neurological condition that, in the opinion of the researcher, could contribute to the subject's cognitive impairment (for example, substances abuse, vitamin B12 deficiency, abnormal thyroid function, stroke, or other Cerebral vascular disease, Lewy body dementia, frontotemporal dementia, TBI).
* A clinically significant psychiatric illness (eg, major depression, schizophrenia, or bipolar affective disorder) in the 6 months prior to screening.
* Transient ischemic attack or cerebrovascular accident or any unexplained loss of consciousness in 1 year before selection (in case of vascular deficit with cognitive sequelae that may still be reversible).
* Poorly controlled diabetes mellitus, due to a glycosylated haemoglobin (HbA1c) value of 8% in the selection.
* History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class 3 or 4), or clinically significant conduction disorders (unstable atrial fibrillation) within 1 year prior to screening.
* Uncontrolled hypertension defined as the mean of 3 measures of systolic blood pressure / diastolic blood pressure> 165/100 mmHg, and persistent systolic blood pressure / diastolic blood pressure > 180/100 mmHg in the 3 months prior to randomization which were considered by the researcher as an indicative of chronic uncontrolled hypertension.
* History of seizures in the 10 years prior the selection.
* Recent history (within 1 year of screening) of alcohol or substance abuse with positive urine test (looking for non-prescription drugs), alcohol or cannabinoids.
* Patients with chronic diseases will be excluded: severe psychiatric, chronic processes in need of treatment such as chronic kidney failure, chronic liver disease, neoplasms under treatment, chronic obstructive pulmonary disease, endocrinopathies susceptible to decompensation and digestive tract diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Cognitive change | Baseline and 24 weeks after each dietary intervention
  Cognitive change in Alzheimer's Disease Assessment Scale-Cognitive-Plus ("ADAS-Cog- Plus"). The total ADAS-Cog-plus score ranges from 0-70 with higher scores suggesting greater impairment.

SECONDARY OUTCOMES:
Microbiota pattern | Baseline and 24 weeks after each dietary intervention
  Changes in the percentage of different families of Microbiota will be analysed during the study
Endotoxemia levels | Baseline and 24 weeks after each dietary intervention
  Changes in the endotoxemia levels will be analysed during the study
Change in inflammatory marker | Baseline and 24 weeks after each dietary intervention
  At time 0 and after 24 weeks of each intervention period and follow-up, the levels of high sesitivity C-reactive protein (hs-CRP) were determined in plasma in mg/dL.
Change in oxidative stress parameters | Baseline and 24 weeks after each dietary intervention
  At time 0 and after 24 weeks of each intervention period and follow-up, the levels of advanced glycation end products (AGEs) were determined in serum in ug/mL: methylglioxal (MG) and N-carboxymethyllysine (CML). Likewise, carbonilated proteins in nmol/mg and lipid peroxidation levels in plasma in ug/mL.
Neurofunctional change | Baseline and 24 weeks after each dietary intervention
  At time 0 and after 24 weeks of each intervention period and follow-up, neurofunctional changes were measured by emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose (18F-FDG-PET)
Modulation of Microbiota-gut-nervous system | Baseline and 24 weeks after each dietary intervention
  Changes in the plasma levels of molecules with activity on the nervous system were analysed during the study. At time 0 and after 24 weeks of each intervention period and follow-up, Gamma-Aminobutiric acid (GABA) in ng/mL and short-chain fatty acids (acetate, propionate and butirate) in ng/mL were determined in plasma.
Change in cytokine levels | Baseline and 24 weeks after each dietary intervention
  At time 0 and after 24 weeks of each intervention period and follow-up, the levels of interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-a) were determined in plasma in pg/mL.
Neuropeptides modulation | Baseline and 24 weeks after each dietary intervention
  Changes in the plasma levels of molecules with activity on the nervous system were analysed during the study. At time 0 and after 24 weeks of each intervention period and follow-up, Substance P (SP), Y Peptide (PYY), beta-amyloid in pg/mL were determined in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Perez-Martinez, PhD, MD, Principal Investigator — IMIBIC/ Reina Sofia University Hospital / University of Cordoba
Locations (1):
- Reina Sofia University Hospital, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cardelo MP, Corina A, Leon-Acuna A, Quintana-Navarro GM, Alcala-Diaz JF, Rangel-Zuniga OA, Camargo A, Conde-Gavilan C, Carmona-Medialdea C, Vallejo-Casas JA, Carmona-Asenjo E, Ochoa-Sepulveda JJ, Aguera-Morales E, Delgado-Lista J, Katsiki N, Lopez-Miranda J, Perez-Jimenez F, Yubero-Serrano EM, Perez-Martinez P. Effect of the Mediterranean diet and probiotic supplementation in the management of mild cognitive impairment: Rationale, methods, and baseline characteristics. Front Nutr. 2022 Dec 8;9:1037842. doi: 10.3389/fnut.2022.1037842. eCollection 2022. PMID 36570150